CLINICAL TRIAL: NCT03696836
Title: Treatment of Medial Knee Joint Pain With the Trammpolin® Meniscus Prosthesis
Brief Title: AIR (Artificial Implant for Medial Meniscus Replacement) Study
Acronym: AIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely
Sponsor: ATRO Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-001
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Meniscectomy; Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trammpolin® meniscus prosthesis (Experimental): The patients will be implanted with the Trammpolin® meniscus prosthesis
  Interventions: Device: Trammpolin® meniscus prosthesis

INTERVENTIONS:
Device: Trammpolin® meniscus prosthesis — Trammpolin® meniscus prosthesis is an anatomically shaped, synthetic medial meniscus replacement

SUMMARY:
The AIR Study is a multi-center, prospective, interventional clinical trial with the objective to evaluate the safety and performance of the Trammpolin® meniscus prosthesis system.

DETAILED DESCRIPTION:
The Trammpolin® meniscus prosthesis is intended to replace the native medial meniscus to provide pain relief in the medial compartment of the knee joint, when this is caused by medial partial meniscectomy.

Patients who meet the inclusion/exclusion criteria and who are implanted with the Trammpolin® meniscus prosthesis will be followed for 2 years. The patient reported outcome measures for knee pain and function, and knee clinical condition by MRI and X-ray is assessed post-operative compared to pre-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Has medial compartment joint pain with > 6 months ago a medial partial meniscectomy as confirmed by patient history and MRI
2. Has a KOOS Pain of ≤ 75 (100 being no pain and the highest attainable score)
3. Is between age 30 and 65 years (inclusive) at the time of screening
4. Has neutral alignment ± 5° of the mechanical axis, i.e., the angle formed by a line drawn from the center of the femoral head to the medial tibial spine and a line drawn from the medial tibial spine to the center of the ankle joint, as confirmed by X-ray
5. Is willing to be implanted with the Trammpolin® meniscus prosthesis.
6. Is able to do the study required follow up visits, questionnaires, X-rays, CT-scans, and MRI's
7. Is able and willing to understand and sign the study Informed Consent Form
8. Is able to read and understand the national language of the country in which the relevant clinical site is located

Exclusion Criteria:

1. Has a symptomatic knee because of a tear that could be addressed by a repeat partial meniscectomy
2. Has evidence of a modified Outerbridge Grade IV cartilage loss on the medial tibial plateau or femoral condyle that potentially could contact a Trammpolin® meniscus prosthesis (e.g., a focal lesion > 0.5 cm2 correlating to a circular defect of > 8 mm in diameter)
3. Has lateral compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the lateral compartment
4. Has a varus or valgus knee deformity of > 5° requiring a tibial or femoral osteotomy
5. Has a varus alignment that is not passively correctable
6. Has a laxity level of more than Grade II (IKDC), primary or secondary to an injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL)
7. Has significant trochlear dysplasia, patellar instability or symptomatic patellar misalignment
8. Has patellar compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the patellar compartment.
9. Compared to a normal knee, has obvious radiological evidence of medial femoral squaring, anatomical variance in the medial tibial plateau, or irregularly shaped cartilage surface
10. Had an ACL reconstruction performed < 9 months prior to surgery
11. Has a BMI > 32.5 at the time of screening
12. Received any type of prosthetic knee implant made of artificial non-resorbable plastic, metal or ceramic, not including the Trammpolin® meniscus prosthesis
13. Has a knee flexion contracture > 10°
14. Has flexion < 90°
15. Had a previous medial femoral condyle surgery (not including microfracture) or High Tibial Osteotomy (HTO)
16. Has insufficiency fractures or avascular necrosis of the medial compartment
17. Has an active infection or tumor (local or systemic)
18. Has any type of knee joint inflammatory disease including Sjogren's syndrome
19. Has neuropathic knee osteoarthropathy, also known as Charcot joint
20. Has any medical condition that does not allow possible arthroscopy of the knee
21. Has neurological deficit (sensory, motor, or reflex)
22. Is currently involved in another investigation of the lower extremity
23. Anticipates having another lower extremity surgery during the study period
24. Is contraindicated for corticosteroid injections (i.e., patients with allergy to any of the components or with idiopathic thrombocytopenic purpura)
25. Has received any corticosteroid knee injections ≤ 3 months prior to surgery
26. Has chondrocalcinosis
27. Has proven osteoporosis
28. Is on immunostimulating or immunosuppressing agents
29. Has ipsilateral or contralateral lower limb joint conditions that may affect ambulation or KOOS (e.g. have a leg length discrepancy > 2.5 cm [1 inch], causing a noticeable limp)
30. Is a female who is lactating, expecting, or is intending to become pregnant during the study period
31. Is an active smoker
32. Is mentally incapacitated (incapable of appraising or controlling conduct) or have mental disability (e.g., dementia or Alzheimer's)
33. Is a prisoner
34. Has a condition or be in a situation that, in the Investigator's opinion, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain sub-scale | 24 Months
  Performance of the Trammpolin® meniscus prosthesis in improving pain
Trammpolin® meniscus prosthesis device related complications | 24 Months
  The nature and frequency of all adverse events observed during the study

SECONDARY OUTCOMES:
KOOS Pain sub-scale | 6 Weeks; 3, 6 and 12 Months
  KOOS Pain sub-scale
Overall KOOS scale | 6 Weeks; 3, 6, 12 and 24 Months
  Overall KOOS scale
Lysholm scale | 6 Weeks; 3, 6, 12 and 24 Months
  Lysholm scale
IKDC objective scale | 6 Weeks; 3, 6, 12 and 24 Months
  IKDC objective scale
Knee X-ray | 6 Weeks; 12 and 24 Months
  Joint space measurement
Knee MRI | 12 and 24 Months
  Cartilage damage and extrusion

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Maastricht UMC+, Maastricht
  - Radboud UMC, Nijmegen
  - Sint Maartenskliniek, Ubbergen

IPD SHARING:
Plan to Share IPD: No